CLINICAL TRIAL: NCT02925975
Title: Early Precise Diagnosis and Intervention of Cirrhotic Portal Hypertension (CPT) Based on a Noninvasive 3D-virtual-model of Hepatic Portal System (3D-vHPS)
Brief Title: Early Precise Diagnosis and Intervention of CPT Based on a Noninvasive 3D-vHPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Changqing Yang (Other)
Collaborators: Shanghai Changzheng Hospital (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Changqing Yang, Chief physician in Digestive department, Professor in Hepatology, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Yang-20161003
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Portal Hypertension; Cirrhosis
MeSH Terms: conditions — Hypertension, Portal; Fibrosis | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Healthy controls (Other): Healthy volunteers are enrolled as controls to get a normal range of pressure gradient in different sites of hepatic portal system (HPS), such as portal vein, superior mesenteric vein, inferior mesenteric vein and splenic vein. All enrolled healthy subjects should undergo anatomic computed tomographic angiography (CTA) and Doppler ultrasound for only one time, to rebuild a 3D-vHPS by computer.
  Interventions: Device: 3D-vHPS
- Treatment group guided by vPVPG (Experimental): Enrolled cirrhotic patients with virtual portal vein pressure gradient (vPVPG) above 12mmHg are only treated by oral carvedilol. Once there are visible varies under the endoscopy, participants will be treated with routine endoscopic procedures.
  Interventions: Drug: Carvedilol; Device: 3D-vHPS; Procedure: Routine endoscopic procedures
- Follow-up group guided by vPVPG (Experimental): Cirrhotic patients with vPVPG lower than 12mmHg are followed-up with anatomic CTA and Doppler ultrasound every six months. Once vPVPG is higher 12mmHg or visible varies under the endoscopy, participants will be rescheduled to treatment group guided by vPVPG.
  Interventions: Drug: Carvedilol; Device: 3D-vHPS
- Follow-up group guided by endoscopy (Active Comparator): Cirrhotic patients are followed-up by routine endoscopy. Once there are visible varies, participants will be treated according to Baveno V consensus in portal hypertension, such as oral carvedilol and routine endoscopic procedures.
  Interventions: Drug: Carvedilol; Device: 3D-vHPS; Procedure: Routine endoscopic procedures

INTERVENTIONS:
Drug: Carvedilol — Carvedilol starts from 6.25mg daily and increase to 12.5mg once daily in next week if being tolerated.
  Other Names: Coreg
  Arms: Follow-up group guided by endoscopy; Follow-up group guided by vPVPG; Treatment group guided by vPVPG
Device: 3D-vHPS — This 3D model of HPS is rebuilt by a software combining the anatomic information of vessels from CTA (computed tomographic angiography) and the blood stream speed of targeted vessel from Doppler Ultrasound.
Procedure: Routine endoscopic procedures — These include esophageal band ligation and tissue glue injection in the fundus of stomach by upper GI endoscopy if there are visible varies in cirrhotic patients. There routine procedures are done to prevent potential varies associated bleeding.
  Arms: Follow-up group guided by endoscopy; Treatment group guided by vPVPG

SUMMARY:
The aim of this study is to investigate the possibilities of early and precise management to decrease portal vein pressure in cirrhotic patients, guided by a non-invasive 3D-virtual-model of hepatic portal system (3D-vHPS). Healthy volunteers are enrolled to determine the normal range of pressure density in different sites of HPS. Cirrhotic patients without visible gastro-esophageal varies by endoscopy are randomly enrolled to virtual portal vein pressure gradient (vPVPG) monitored or non-vPVPG monitored groups. Non-vPVPG groups are followed-up and treated according to Baveno V consensus in portal hypertension. Patients in vPVPG-monitored groups are followed-up by anatomic computed tomographic angiography (CTA) and Doppler ultrasound every six months. Once vPVPG is above 12mm of mercury (Hg), participants will receive carvedilol treatment. All cirrhotic patients are followed-up with the incidence of portal hypertension-related complications, mortality rate and life quality assessment.

DETAILED DESCRIPTION:
The non-invasive 3D-HPS is a newly-developed test to determine vPVPG based on anatomic computed tomographic angiography (CTA) and Doppler ultrasound. In this study, vPVPG is determined by the 3D-HPS.

ELIGIBILITY:
Inclusion Criteria:

* Proven cirrhosis based on histology or unequivocal clinical, sonographic and laboratory findings
* Child-Pugh score < 9
* No visible gastro-esophageal varies by endoscopy

Exclusion Criteria:

* Patients with malignant diseases
* Treatment with vasoactive drugs
* Prior transjugular intrahepatic portosystemic stent-shunt surgery
* Patients with known allergy to iodinated contrast
* Treatment with immunosuppressants
* Renal sufficiency
* Patients with coronary artery diseases, or treated with anticoagulants
* Pregnancy
* Inability to adhere the follow-up
* Any life-threatening disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of portal hypertensive complications: ascites and variceal bleeding | 3 years
10% decrease of virtual hepatic venous pressure gradient (HVPG) from baseline level | 3 years

SECONDARY OUTCOMES:
Mortality rate | 3 years

OTHER OUTCOMES:
Quality of life | 3 years
  The short form Health Survey (SF36-V2)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided